CLINICAL TRIAL: NCT05136313
Title: Healthy vs Unhealthy Obesity in Young Male Adults: Early Predictors, Mechanistic Insights and Effects of Time-Restricted Eating
Brief Title: Healthy vs Unhealthy Obesity: Mehanistic Insights and Effects of Time-Restricted Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Nutrición y Tecnología de los Alimentos (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other); Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Mariana Cifuentes, Professor, Instituto de Nutrición y Tecnología de los Alimentos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1211477
Record Dates: First submitted 2021-11-17; First posted 2021-11-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Metabolically Healthy Obesity; Intermittent Fasting
Keywords: Time restricted eating; Metabolic health; PBMC; Adipokines
MeSH Terms: conditions — Obesity, Metabolically Benign; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: TRE intervention comparing MHO vs MUO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHO (Experimental): metabolically healthy obese subjects undergoing TRE
  Interventions: Behavioral: Time-restricted eating
- MUO (Experimental): metabolically unhealthy obese subjects undergoing TRE
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — 16 weeks of TRE consisting of an 8-hour eating window.
  Other Names: Time-restricted feeding; Intermittent fasting

SUMMARY:
Obesity-related cardiometabolic diseases are now a leading cause of death worldwide. These diseases result from a dysfunctional adipose tissue (AT) that induces inflammation, insulin resistance and altered endocrine function. However, not all obese people develop metabolic complications, which has given rise to the concept of "metabolically healthy obesity" (MHO). Recent evidence suggests that intermittent fasting methods, in particular time-restricted eating (TRE) may be effective in improving cardiometabolic health, independently of weight loss, and this could be particularly effective in MUO subjects. The investigators hypothesize that in young male adults TRE is a more effective/beneficial approach in MUO than in MHO due to the weight loss-independent improvement in their inflammatory and metabolic derangements. To this aim, a 16-week 8h TRE intervention study will be performed in MHO and MUO subjects, assessing anthropometric, endocrine, and other outcomes.

DETAILED DESCRIPTION:
Although clinical differences between metabolically healthy and unhealthy obesity (MHO and MUO, respectively) have been extensively described, cellular mechanisms involved in these different phenotypes are largely unknown. This evidence is crucial for proposing preventive and therapeutic approaches. Recently, intermittent fasting methods, in particular time-restricted eating (TRE, a self-selected daily limited eating window protocol), have shown to be effective in improving cardiometabolic health, independently of weight loss, which could be particularly relevant in MUO.

The investigators will recruit young (20-22y-old) males with obesity (Body Mass Index≥30) and classify them as MHO or MUO (≤1 or ≥3 metabolic syndrome risk factors, respectively). A 16-week, 8h TRE intervention will be conducted in MHO vs. MUO subgroups, to assess and compare the anthropometric, metabolic, endocrine, inflammatory and peripheral blood mononuclear cell (PBMC) mechanistic/signaling response.

The investigators expect to advance the understanding of cellular mechanisms implicated in MHO and MUO, including potential therapeutic targets. Ultimately, the investigators expect to find relevant opportunities for intervention to prevent the serious cardiometabolic consequences of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Belong to the GOCS cohort at INTA
* BMI≥30
* Own and use a Smartphone with Apple iOS or Android OS
* Baseline eating period ≥ 13 h per day.

Exclusion Criteria:

* Medications for any metabolic syndrome disorder
* Shift workers
* Known inflammatory and/or rheumatologic disease
* History of cardiovascular event
* Thyroid or adrenal disease, malignancy or diabetes
* History of eating disorder.
* Special diet (e.g., celiac disease),or any other disease or treatment that may interfere with the study.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
TG | 16 weeks
  Fasting triglycerides

SECONDARY OUTCOMES:
Waist circumference | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Cifuentes, PhD, Principal Investigator — Universidad de Chile INTA
Locations (1):
- INTA, Universidad de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Undecided